CLINICAL TRIAL: NCT05774626
Title: Continuation of Subcutaneous and Intramuscular Injectable Contraception: a Non-randomized Prospective Cohort Study in Punjab, Pakistan
Brief Title: Injectable Contraception Cohort Study in Punjab, Pakistan
Status: Completed | Type: Observational
Sponsor: Jhpiego (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00021562
Record Dates: First submitted 2022-11-28; First posted 2023-03-17 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Contraceptive Usage
Keywords: injectable contraception; prospective cohort study; Pakistan
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DMPA-SC: All married women of reproductive age who receive family planning counseling at a participating health facility and who choose to receive injectable contraception will be given an option of either DMPA-IM (current health worker administered standard of care) or DMPA-SC (new administration method, with option for self-injection after completing training). Those opting for DMPA-SC will receive training on self-injection procedures and an opportunity to practice injection procedures on a model (e.g. condom filled with salt) to demonstrate confidence and proficiency to inject herself under the supervision of a healthcare provider. Clients will then be shown how to use a calendar to determine when their next injection is due, and provided a calendar/reminder card, job aids that illustrate self-injection steps (including safe disposal of needles), and 3 doses of DMPA-SC to take home for future use.
  Interventions: Behavioral: Contraceptive usage
- DMPA-IM: All married women of reproductive age who receive family planning counseling at a participating health facility and who choose to receive injectable contraception will be given an option of either DMPA-IM (current health worker administered standard of care) or DMPA-SC (new administration method, with option for self-injection after completing training).
  Interventions: Behavioral: Contraceptive usage

INTERVENTIONS:
Behavioral: Contraceptive usage — Continued use of injectable contraception, administered on a quarterly basis

SUMMARY:
The aim of this study is to assess the value proposition of expanding contraceptive options available to women in Punjab, Pakistan to include subcutaneous depot medroxyprogesterone acetate (DMPA-SC).

Specific objectives are:

1. To compare 12-month continuation rates for DMPA-SC and intramuscular DMPA (DMPA-IM) among married women 18- 49 years of age in two districts of Punjab, Pakistan
2. To understand how characteristics and experiences of DMPA-SC and DMPA-IM users differ.
3. To assess how well women opting for self-injection of DMPA-SC adhere to standards for commodity storage, injection timing, injection technique, and waste disposal

DETAILED DESCRIPTION:
Depot medroxyprogesterone acetate (DMPA) is a highly-effective, injectable contraceptive method that requires injections every 11 to 17 weeks. It is available in both intramuscular (IM) and subcutaneous (SC) formulations, which are therapeutically equivalent and have similar safety profiles. DMPA-IM has been included in the method mix for most countries for many years. DMPA-SC is a newer formulation being added to the method mix in select settings. Studies demonstrate that self-administration of subcutaneous DMPA (DMPA-SC) outside clinical settings is safe, effective, feasible, acceptable, and can improve continuation, and a recommendation in favor of self-injected DMPA-SC is included in WHO guidelines on self-care interventions for health and well-being.

The Bill and Melinda Gates Foundation is funding implementation research in multiple countries to understand how self-injection of DMPA-SC can best be introduced to specific markets to expand the contraceptive options available to women and girls, health system characteristics, the demand for self-injection when DMPA-SC is offered alongside a range of other methods, and women's and girl's ability to start and continue use. Jhpiego has received funding to conduct one of these 'market tests' in Punjab, Pakistan.

The aim of this study is to assess the value proposition of expanding contraceptive options available to women in Punjab, Pakistan to include subcutaneous depot medroxyprogesterone acetate (DMPA-SC).

Specific objectives are:

1. To compare 12-month continuation rates for DMPA-SC and intramuscular DMPA (DMPA-IM) among married women 18- 49 years of age in two districts of Punjab, Pakistan
2. To understand how characteristics and experiences of DMPA-SC and DMPA-IM users differ.
3. To assess how well women opting for self-injection of DMPA-SC adhere to standards for commodity storage, injection timing, injection technique, and waste disposal

ELIGIBILITY:
Inclusion Criteria:

* Married women aged 18-49 years
* Decide to use injectable contraception and meet WHO medical eligibility criteria for injectable use
* Want to avoid pregnancy for at least 12 months
* Live within study districts
* Are willing to be contacted by study team members via telephone and/or in-person

Exclusion Criteria:

* Women under age 18 and above 49
* Unmarried women
* Hope to become pregnant within next 12 months
* Do not reside within study districts
* Are not willing to be contacted by study team members via telephone or in-person
* Lack cognitive capacity to give informed consent or complete interviews

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Clients receiving family planning counseling and services at participating public and private health facilities in Kasur and Khanewal districts of Punjab, Pakistan
Sampling Method: Non-Probability Sample
Enrollment: 1009 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
DMPA continuation rate | up to 12 months
  Participant use of DMPA measured at 3, 6 and 9 months following enrollment (providing coverage for 3 months with each dose)

OTHER OUTCOMES:
Characteristics of women in the two study groups (DMPA-SC and DMPA-IM users) | At enrollment
  Demographics, contraceptive history, decision-making, reasons for choosing method, reproductive empowerment, self-confidence
Family planning service provision and injectable contraceptive use experiences of women in the two study groups (DMPA-SC and DMPA-IM users) | Up to 12 months
  Experiences receiving family planning services and with chosen contraceptive method

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Tappis, DrPH, Principal Investigator — Jhpiego
Locations (41):
- Pakistan (41):
  - Bhu 76/10-R, Khanewal, Pubjab
  - BHU Fatehpur, Kasur, Punjab Province
  - BHU Herdo Sehari, Kasur, Punjab Province
  - BHU Pakhoki, Kasur, Punjab Province
  - BHU Rao Khan Wala, Kasur, Punjab Province
  - BHU Serhali, Kasur, Punjab Province
  - BHU Sheikh Bhago, Kasur, Punjab Province
  - Fatima Maternity Home, Kasur, Punjab Province
  - FHC Kasur, Kasur, Punjab Province
  - FWC Chunian-1, Kasur, Punjab Province
  - FWC Kasur 5, Kasur, Punjab Province
  - FWC Kotha Kalan, Kasur, Punjab Province
  - FWC Qaiser Garh, Kasur, Punjab Province
  - FWC Rosa Tibba, Kasur, Punjab Province
  - FWC Sheikh Umad Kohna, Kasur, Punjab Province
  - FWC Talwandi, Kasur, Punjab Province
  - Hajra Maternity Home, Kasur, Punjab Province
  - Rafique Maternity Home, Kasur, Punjab Province
  - RHC Changamanga, Kasur, Punjab Province
  - RHC Ellabad, Kasur, Punjab Province
  - RHC Gandasingh, Kasur, Punjab Province
  - RHC Khuddian, Kasur, Punjab Province
  - RHC Mustafabad, Kasur, Punjab Province
  - Ali Maternity Home, Khanewal, Punjab Province
  - Bhu 171/10-R, Khanewal, Punjab Province
  - Bhu 30/10-R, Khanewal, Punjab Province
  - Bhu 44/15-L, Khanewal, Punjab Province
  - Bhu 79/10-R, Khanewal, Punjab Province
  - Bhu 92/10-R, Khanewal, Punjab Province
  - Bhu 92/15-L, Khanewal, Punjab Province
  - BHU Chack 131/15 L, Khanewal, Punjab Province
  - FHC DHQ Khanewal, Khanewal, Punjab Province
  - FHC THQ Mian Cahnu, Khanewal, Punjab Province
  - FWC Kacha Khuh, Khanewal, Punjab Province
  - FWC Makhdoom Pur, Khanewal, Punjab Province
  - FWC Model Center, Khanewal, Punjab Province
  - RHC Kacha Khuh, Khanewal, Punjab Province
  - RHC Makhdom pur, Khanewal, Punjab Province
  - RHC Tulamba, Khanewal, Punjab Province
  - Tehseen Surgical Clinic, Khanewal, Punjab Province
  - Zainab Maternity Home, Khanewal, Punjab Province

IPD SHARING:
Plan to Share IPD: No
A deidentified analytical dataset will be posted in an open access repository upon study completion.

REFERENCES:
- [Derived] Tappis H, Qayyum K, Bryce E, Fatima A, Christofield M, Haider H, Ameen A, Gardezi SMA, Rafay F, Assad F. Injectable contraceptive continuation and user experiences in Punjab, Pakistan: a non-randomized prospective cohort study protocol. BMC Womens Health. 2025 Sep 7;25(Suppl 1):427. doi: 10.1186/s12905-025-03969-9. PMID 40916043